CLINICAL TRIAL: NCT06482125
Title: Emergence Agitation in Pediatrics After Dexmedetomidine vs. Sevoflurane Anesthesia: a Randomized Controlled Trial
Brief Title: Emergence Agitation Between Dexmedetomidine and Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pelita Harapan University (Other)
Responsible Party: Principal Investigator, Corry Quando Yahya, Pediatric Anesthesiologist and Lecturer at Pelita Harapan University, Department of Anesthesia and Intensive Care, Pelita Harapan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 183/K-LKJ/ETIK/V/2024
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Emergence Delirium
Keywords: Emergence Agitation; Dexmedetomidine; Delirium; Children; Facial Cleft
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Dexmedetomidine; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Pediatrics ages 3 months to 10 years
Who Masked: Participant
Masking Description: Patients are selected randomly using a computer-generated device to become a control arm or a treatment arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalation Sevoflurane (Active Comparator): Participants in this group will receive inhalation anesthesia Sevoflurane at 2-3 Vol% as their sole anesthetic maintenance agent throughout the surgical procedure.
  Interventions: Drug: Sevoflurane
- Total Intravenous Dexmedetomidine (Experimental): Participants in this group will receive Total Intravenous Dexmedetomidine as their sole anesthetic maintenance agent. Intravenous Dexmedetomidine 1.5ug/kg will be administered within 10 minutes and maintenance dose of 1.5ug/kg/hour will be given throughout the surgical procedure.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intervention group will receive Total Intravenous Dexmedetomidine as their anesthetic maintenance agent. Intravenous Dexmedetomidine 1.5ug/kg will be administered within 10 minutes and maintenance dose of 1.5ug/kg/hour continued as the sole anesthetic maintenance agent, thereafter.
  Other Names: Intravenous Dexmedetomidine
  Arms: Total Intravenous Dexmedetomidine
Drug: Sevoflurane — Inhalation Sevoflurane will be administered as an anesthetic maintenance agent. Sevoflurane at 2 - 3 Vol% will be administered throughout the operative procedure.
  Other Names: Inhalation Sevoflurane
  Arms: Inhalation Sevoflurane

SUMMARY:
Emergence agitation is commonly encountered after receiving inhalation anesthesia. This distressing phenomenon carries risks that are harmful to patients, caregivers and medical personnel. Using total intravenous Dexmedetomidine, the investigators seek to reduce agitation and provide gentle emergence from anesthesia.

DETAILED DESCRIPTION:
Surgery for pediatric cleft lip and palate repair often utilizes high dose opioids and inhaled anaesthesia, thereby causing postoperative complications such as desaturation and/or severe agitation after anesthesia. These complications are detrimental to the child, medical personnel and causes tremendous psychologic stress to parents. This study aims to decrease these complications through Dexmedetomidine, an Alpha-2 receptor agonist with anxiolytic, sympatholytic and analgetic properties. Devoid of respiratory depressant effect, it allows patients to maintain effective ventilation and reduce agitation, postoperatively. Its unique anesthetic property may shed light to provide safe anesthesia and gentle emergence to this young, vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with weight ranging 5 kg - 25 kg
2. Patients with American Society of Anesthesiologist (ASA) Physical Status Classification 1 and 2

Exclusion Criteria:

1. Patients with any acquired congenital syndrome
2. Patients who are actively taking anti-seizure medications and/or has been diagnosed with epilepsy
3. Patients with functional and structural abnormalities of the heart, including arrythmias
4. Patients with liver disease

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hori Hariyanto, MD, Study Director — Pelita Harapan University
Locations (1):
- Pelita Harapan University, Tangerang, Banten, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data and other supporting information will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 31 July 2024 up to 31 December 2024
Access Criteria: Data may be accessed for audit purposes

REFERENCES:
- [Result] Liu D, Pan L, Gao Y, Liu J, Li F, Li X, Quan J, Huang C, Lian C. Efficaciousness of dexmedetomidine in children undergoing cleft lip and palate repair: a systematic review and meta-analysis. BMJ Open. 2021 Aug 16;11(8):e046798. doi: 10.1136/bmjopen-2020-046798. PMID 34400450
- [Result] Peng W, Zhang T. Dexmedetomidine decreases the emergence agitation in infant patients undergoing cleft palate repair surgery after general anesthesia. BMC Anesthesiol. 2015 Oct 13;15:145. doi: 10.1186/s12871-015-0124-7. PMID 26464000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria were: American Society of Anesthesiologists (ASA) physical status I or II patients, weighing not more than 25 kg were scheduled to undergo cleft lip or palate repair.
  Exclusion criteria were children with congenital heart disease; syndromic children, and/or children with a history of epilepsy and liver dysfunction.
Groups:
- Inhalation Sevoflurane: Participants in this group will receive inhalation anesthesia Sevoflurane at 2-3 Vol% as their sole anesthetic maintenance agent throughout the surgical procedure.
  Inhalation Sevoflurane: Inhalation Sevoflurane will be administered as an anesthetic maintenance agent. Sevoflurane at 2 - 3 Vol% will be administered throughout the operative procedure.
- Total Intravenous Dexmedetomidine: Participants in this group will receive Total Intravenous Dexmedetomidine as their sole anesthetic maintenance agent. Intravenous Dexmedetomidine 1.5ug/kg will be administered within 10 minutes and maintenance dose of 1.5ug/kg/hour will be given throughout the surgical procedure.
  Total Intravenous Dexmedetomidine: Intervention group will receive Total Intravenous Dexmedetomidine as their anesthetic maintenance agent. Intravenous Dexmedetomidine 1.5ug/kg will be administered within 10 minutes and maintenance dose of 1.5ug/kg/hour continued as the sole anesthetic maintenance agent, thereafter.
Period: Overall Study
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine
Started (July 31, 2024) | 62 | 59
Completed (December 31, 2024) | 62 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inhalation Sevoflurane: Subjects receiving Sevoflurane as their maintenance anesthetic
- Total Intravenous Dexmedetomidine: Subjects receiving Dexmedetomidine as their maintenance anesthetic
- Total: Total of all reporting groups
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Continuous [Median (Full Range); unit: months] — Age is measured from the subject's birth date up to the date of surgery (in months).
  months | 24 [3 to 120] | 24 [3 to 120] | 24 [3 to 120]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 62 | 59 | 121
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight (kg) [Mean (Standard Deviation); unit: kilogram] | 11.4 (5.4) | 10.6 (5.0) | 10.9 (5.2)
Type of operation (Labioplasty/Palatoplasty) [Count of Participants; unit: Participants]
  Labioplasty | 30 | 33 | 63
  Palatoplasty | 32 | 26 | 58
Preschool Children [Mean (Standard Deviation); unit: years] — Ages Two to Five years old Population: Measures preschool children ages only 2 to 5 years old, population at high risk to experience emergence agitation
  years
    number analyzed (Participants) | 21 | 21 | 42
    (all) | 3.4 (1.1) | 3.2 (1.1) | 3.3 (1.1)
Modified Yale Preoperative Anxiety Scale (mYPAS) [Mean (Standard Deviation); unit: units on a scale] — Patients were assessed at the preoperative clinic one day before their surgery. mYPAS is an observational instrument that covers 4 items is the current "criterion standard" for assessing child anxiety.
  Scoring: The mYPAS produces 4 scores, 1 score for each of the 4 behaviors. Each score is calculated by dividing each item rating by the highest possible rating (i.e., 6 for the "vocalizations" item and 4 for all other items), adding all the produced values, dividing by 4, and multiplying by 100. Minimum score is 22.75, maximum is 100 (< 30 is anxious, > or equal 30 is not anxious). Population: Only measures Preschool children population ages 2 - 5 years old
  units on a scale
    number analyzed (Participants) | 21 | 21 | 42
    (all) | 56.1 (13.7) | 54.3 (15.0) | 55.2 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Emergence Agitation
Description: Cravero scale uses a numeric scale. 1 = obtunded with no response to stimulation; 2 = asleep, but responsive to movement or stimuli; 3 = awake and responsive, 4 = crying; 5 = thrashing behavior that requires restraint. Minimum values of NOT AGITATED is 1.0 up to maximum of 2.9. Minimum values of AGITATED is 3.10 up to maximum of 5.0. Cravero scale is measured from the moment of extubation and every 15 minutes thereafter until the patient is completely awakened (in the recovery room). The total score is summed, and the average is reported.
Time Frame: Assessed starting the time of extubation and every 15 minutes interval until the patient is completely awake in the recovery room. The average of all values throughout the observation period was summed and the average scale reported.
Population: Scale of 1.0 - 2.9 indicates no emergence agitation, a scale of 3.0 - 5.0 indicates emergence agitation
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Inhalation Sevoflurane; Total Intravenous Dexmedetomidine: Cravero Score is measured every 15 minutes until patient has fully recovered. The average score per person is reported.
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine
Number analyzed (Participants) | 62 | 59
Score on a scale | 3.9 (0.9) | 2.5 (0.6)
Statistical Analysis 1: Comparison: Inhalation Sevoflurane vs Total Intravenous Dexmedetomidine; Test type: Superiority; p = 0.001, Chi-squared, Corrected; Odds Ratio (OR) = 40.955, 95% CI 2-sided [14.098 to 118.972]

2. Primary Outcome: Duration of Anesthesia (Minutes)
Description: Measures the time of anesthesia (in minutes) starting from induction of anesthesia to the termination of anesthetic agent
Time Frame: From time of anesthesia induction up to the termination of anesthetic agent, assessed up to two hours.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Inhalation Sevoflurane: Subject receiving Sevoflurane as their anesthetic maintenance agent.
- Total Intravenous Dexmedetomidine: Subjects receiving Dexmedetomidine as their anesthetic maintenance agent
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine
Number analyzed (Participants) | 62 | 59
minutes | 50 (17) | 46 (15)
Statistical Analysis 1: Comparison: Inhalation Sevoflurane vs Total Intravenous Dexmedetomidine; Test type: Equivalence — The threshold for statistical significance is p < 0.05; p = 0.345, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Duration of Surgery (Minutes)
Description: Measures the time of surgery after the application of sterile draping up to the end of surgery.
Time Frame: From time of surgery up to the termination of anesthetic agent, assessed up to two hours.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Inhalation Sevoflurane: Subjects receiving inhalation Sevoflurane as their anesthetic maintenance agent
- Total Intravenous Dexmedetomidine: Subjects receiving intravenous Dexmedetomidine as their anesthetic maintenance agent
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine
Number analyzed (Participants) | 62 | 59
minutes | 41 (15) | 39 (14)
Statistical Analysis 1: Comparison: Inhalation Sevoflurane vs Total Intravenous Dexmedetomidine; Test type: Equivalence — The threshold for statistical significance is p < 0.05; p = 0.450, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time to Extubation (Minutes)
Description: Measures the amount of time taken to extubate. Time is recorded from the moment Sevoflurane is stopped or Dexmedetomidine infusion is stopped until the patient is fit to extubated.
Time Frame: Maximum time to extubate was up to 26 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Inhalation Sevoflurane; Total Intravenous Dexmedetomidine: Time to extubation is recorded in minutes
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine
Number analyzed (Participants) | 62 | 59
minutes | 9.5 (3.7) | 10.4 (4.6)
Statistical Analysis 1: Comparison: Inhalation Sevoflurane vs Total Intravenous Dexmedetomidine; Test type: Equivalence — Reject H0 = the means are equivalent; p = 0.356, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1.00

5. Secondary Outcome: Time to Full Recovery
Description: Measures amount of time taken to full awakening. Time is recorded from the moment of extubation until patient completely awaken at the recovery room area.
Time Frame: Maximum time observed was up to 105 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Inhalation Sevoflurane; Total Intravenous Dexmedetomidine: Time to full recovery or fully awake is recorded in minutes
Arm/Group | Inhalation Sevoflurane | Total Intravenous Dexmedetomidine
Number analyzed (Participants) | 62 | 59
minutes | 51.7 (16.3) | 59.9 (16.4)
Statistical Analysis 1: Comparison: Inhalation Sevoflurane vs Total Intravenous Dexmedetomidine; Test type: Equivalence — Reject H0 = the means are equivalent; p = 0.07, t-test, 2 sided; Mean Difference (Final Values) = 8.202, 95% CI 2-sided [2.310 to 14.095]

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Inhalation Sevoflurane; Intravenous Dexmedetomidine: Adverse events such as hypotension, bradycardia, cardiac arrest or admission to intensive care unit.
Arm/Group | Inhalation Sevoflurane | Intravenous Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 0/62 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT06482125/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT06482125/ICF_001.pdf